CLINICAL TRIAL: NCT03641040
Title: The Analysis of Ocular Deviations Between Dominant and Non-dominant Eye Using Video-oculography (VOG) in Intermittent Exotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Sung-Hyuk Moon, professor, Inje University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IJ1357913579
Record Dates: First submitted 2018-08-19; First posted 2018-08-21 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Intermittent Exotropia; Strabismus
Keywords: Video-oculography; Intermittent exotropia; ocular deviation
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOG group (Experimental): Measurement: Video-oculography(VOG) measure and analyze angles of ocular deviations between dominant and non-dominant eye using VOG with alternate cover.
  Interventions: Diagnostic Test: Video-oculography
- APCT group (Active Comparator): Measurement: Alternative prism cover test(APCT) measure and analyze angles of ocular deviations between dominant and non-dominant eye using APCT
  Interventions: Diagnostic Test: Alternative prism cover test

INTERVENTIONS:
Diagnostic Test: Video-oculography — measure and analyze angles of ocular deviations between dominant and non-dominant eye using VOG with alternate cover.
  Arms: VOG group
Diagnostic Test: Alternative prism cover test — measure and analyze angles of ocular deviations between dominant and non-dominant eye using APCT
  Arms: APCT group

SUMMARY:
Fifteen subjects with intermittent exotropia were included. The subjects were asked to fixate on a black-on-white optotype at 1 m, which subtended a visual angle of 50 min of arc, equating to a Snellen optotype of 20/200. The video files and data about ocular deviations were obtained using VOG with alternate cover test. Investigators analyzed angles of ocular deviations in dominant and non-dominant eyes, compared with values of VOG and deviation angles of the alternative prism cover test.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity >= 1.0/1.0
* Intermittent exotropia
* Cooperative

Exclusion Criteria:

* Other eye disease
* Have hyperopia, myopia > 2 diopter
* Have horizontal strabismus > 50 prism diopter
* Not cooperative, no agree

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
The angles of ocular deviations between dominant and non-dominant eye using VOG with alternate cover | 2 weeks after approval
  The angles of ocular deviations between dominant and non-dominant eye using VOG with alternate cover

CONTACTS AND LOCATIONS:
Locations (1):
- Busan Paik hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided